CLINICAL TRIAL: NCT02704026
Title: Nutritional Status and Body Composition in Children With Inflammatory Bowel Disease: A Prospective Cohort Study
Brief Title: Nutritional Status and Body Composition in Childhood Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Zarife Kuloglu, Professor (M.D.), Ankara University
Other Study IDs: 15H0230004
Record Dates: First submitted 2016-02-17; First posted 2016-03-09 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2018-01

CONDITIONS: Inflammatory Bowel Disease
Keywords: Body composition; Nutritional status
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Body Composition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Inflammatory Bowel Disease: Patients 6-18 of age at the time of enrolment who have IBD at any stage of disease activity, on any or no treatment
  Interventions: Other: Assesment of nutritional status and body composition
- Control: Age- and sex-matched healthy controls
  Interventions: Other: Assesment of nutritional status and body composition

INTERVENTIONS:
Other: Assesment of nutritional status and body composition — At the time of enrollment and after 1 year, anthropometric measurements and assessment of body composition by bioelectrical impedance will be performed for each child

SUMMARY:
Malnutrition and growth retardation are common in children with inflammatory bowel disease (IBD), especially in Crohn's Disease (CD). Malnutrition is associated with disease type, anatomical location, severity of disease and age of patient. Recently, it is reported that almost all children with CD and half with Ulcerative Colitis (UC) have reduced lean mass, however, body fat alteration are not well defined.

The aim of this prospective and observational study was to evaluate nutritional and growth status and body composition of children with IBD using anthropometric measurement and bioelectrical impedance during 1 year follow-up.

DETAILED DESCRIPTION:
Patients 6 to 18 years of age at the time of enrolment who have IBD at any stage of disease activity, on any or no treatment and age- and sex-matched healthy controls will be included. All participants will be followed for 1 year.

Written informed consent will be obtained from the parents or guardians of the participants at the time of enrolment. Prospective and retrospective data will be collected. Complete family and medical history, physical examination and laboratory findings will be recorded on standard case report form. Disease activity will be scored using the Paediatric Crohn's Disease Activity Index for children with CD and the Pediatric Ulcerative Colitis Activity index for those with UC. Endoscopic data will be reviewed and disease location will be classified according to Paris classification. Puberty will be assessed based on the development of secondary sexual characteristics. At the time of enrollment and after 1 year, anthropometric measurements including height, weight, triceps skin fold thickness, middle arm circumference and assessment of body composition by bioelectrical impedance will be performed for each child. Anthropometric data will be standardized by generation of z-scores for height and weight based on age and gender. Growth deficiency for height and weight measurements will be defined as a z-score\-2.

ELIGIBILITY:
Inclusion Criteria:

* A male or female of 6 to 18 years of age at the time of enrolment
* For children with IBD; the diagnosis of IBD are based on the combination of clinical features and serological, endoscopic, colonoscopic, and histological findings
* For controls : no evidence of inflammatory or chronic disease

Exclusion Criteria:

* A male or female < 6 years or > 18 years old at the enrollment

  * For children with IBD : Presence of other chronic diseases
  * For healthy control: Any coexisting chronic disease known to affect growth, nutritional status, dietary intake, or development

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with IBD at any stage of disease activity, on any or no treatment and age- and sex-matched healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Body mass index | 1 year
  kg/m
Triceps skin fold thickness | 1 year
Middle arm circumference | 1 year
Body composition | 1 year
  fat (%), fat mass and fat-free mass
Paediatric Crohn's Disease Activity Index | 1 year
Paediatric Ulcerative colitis Activity Index | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Zarife Kuloglu, Study Director — Ankara University
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Kugathasan S, Nebel J, Skelton JA, Markowitz J, Keljo D, Rosh J, LeLeiko N, Mack D, Griffiths A, Bousvaros A, Evans J, Mezoff A, Moyer S, Oliva-Hemker M, Otley A, Pfefferkorn M, Crandall W, Wyllie R, Hyams J; Wisconsin Pediatric Inflammatory Bowel Disease Alliance; Pediatric Inflammatory Bowel Disease Collaborative Research Group. Body mass index in children with newly diagnosed inflammatory bowel disease: observations from two multicenter North American inception cohorts. J Pediatr. 2007 Nov;151(5):523-7. doi: 10.1016/j.jpeds.2007.04.004. Epub 2007 Aug 24. PMID 17961699
- [Background] Markowitz J, Grancher K, Rosa J, Aiges H, Daum F. Growth failure in pediatric inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 1993 May;16(4):373-80. doi: 10.1097/00005176-199305000-00005. PMID 8315544
- [Background] Burnham JM, Shults J, Semeao E, Foster BJ, Zemel BS, Stallings VA, Leonard MB. Body-composition alterations consistent with cachexia in children and young adults with Crohn disease. Am J Clin Nutr. 2005 Aug;82(2):413-20. doi: 10.1093/ajcn.82.2.413. PMID 16087987
- [Background] Sylvester FA, Leopold S, Lincoln M, Hyams JS, Griffiths AM, Lerer T. A two-year longitudinal study of persistent lean tissue deficits in children with Crohn's disease. Clin Gastroenterol Hepatol. 2009 Apr;7(4):452-5. doi: 10.1016/j.cgh.2008.12.017. Epub 2008 Dec 27. PMID 19249399
- [Background] Thangarajah D, Hyde MJ, Konteti VK, Santhakumaran S, Frost G, Fell JM. Systematic review: Body composition in children with inflammatory bowel disease. Aliment Pharmacol Ther. 2015 Jul;42(2):142-57. doi: 10.1111/apt.13218. Epub 2015 Jun 4. PMID 26043941